CLINICAL TRIAL: NCT03932513
Title: A Phase 2, Open-label Study Evaluating the Intra-hepatic Effect of Inarigivir 400 mg Per Day and 400 mg Three Times Per Week on Immune Response and Viral Markers in Virally Suppressed Patients With Chronic Hepatitis B Infection
Brief Title: Evaluating the Effects of Inarigivir on Immune Response and Viral Markers in Chronic Hepatitis B Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was halted due to suspected liver injury in another study with Inarigavir
Sponsor: F-star Therapeutics, Inc. (Industry)
Collaborators: CSI Medical Research Pte Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBP-9200-HBV-203
Record Dates: First submitted 2019-03-22; First posted 2019-04-30 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: HBV; Hepatitis B; Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B; Hepatitis B, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A: inarigivir soproxil (Experimental): Inarigivir 400 mg once per day for 6 weeks (2800mg/week).
  Interventions: Drug: inarigivir soproxil
- Treatment B: inarigivir soproxil (Experimental): Inarigivir 400 mg three times per week for 6 weeks (1200mg/week).
  Interventions: Drug: inarigivir soproxil

INTERVENTIONS:
Drug: inarigivir soproxil — Inarigivir 200mg and 400mg oral tablets, once daily
  Other Names: SB 9200

SUMMARY:
A single center, open-label, study to evaluate the intra-hepatic effect of inarigivir dose per day and three times per week on immune response and viral markers in virally suppressed patients with chronic hepatitis B infection

DETAILED DESCRIPTION:
This is a single center, open-label, study to evaluate the intra-hepatic effect of inarigivir dose per day and three times per week on immune response and viral markers in virally suppressed patients with chronic hepatitis B infection

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥ 21 to ≤ 70 years
2. Chronic hepatitis B infection defined as HBsAg positive and on NUC therapy for at least one year.

   1. Have at least one prior documented result of HBV DNA ≤ 20 IU/mL LLOQ from a local laboratory, 6 or more months prior to Screening
   2. HBV DNA ≤ 20 IU/mL at Screening tested by the Central Laboratory
   3. Have been on a commercially available HBV oral antiviral (OAV) treatment(s) (tenofovir alafenamide, tenofovir disoproxil fumarate, entecavir, adefovir, lamivudine, telbivudine, either as single agents or in combination) with no change in regimen for 3 months prior to screening.
3. Ultrasound, computed tomography (CT) scan, or magnetic resonance imaging (MRI) within 3 months of randomization date with no evidence of hepatocellular carcinoma
4. Must be willing and able to comply with all study requirements including two liver biopsies
5. Negative urine or serum pregnancy test (for women of childbearing potential documented within the 24-hour period prior to the first dose of test drug. If the urine pregnancy test is positive, a follow-up serum test is required for confirmation. Additionally, all fertile males with partners of childbearing age and females must be using reliable contraception during the study and for 3 months after treatment completion. All fertile males must also refrain from sperm donation while on Active drug and for 3 months after completion of Active drug.
6. Must have the ability to understand and sign a written informed consent form; consent must be obtained prior to initiation of study procedures

Exclusion Criteria:

1. Any liver biopsy evidence of metavir F3 or F4 disease on any prior biopsy
2. Any history of decompensation of liver disease including history of ascites, encephalopathy, or varices
3. Evidence of advanced fibrosis at screening as defined by Fibroscan at the Screening Visit of ≥ 8 kilopascals
4. Laboratory parameters not within defined thresholds: ALT or AST ≥ 40 IU, white blood cells < 4500 cells/μL (SI unit < 4.5 × 109/L), hemoglobin (HgB) < 12 g/dL (SI unit < 120 g/L) for females, < 13 g/dL (SI unit < 130 g/L) for males, platelets < 150,000 per μL (SI unit < 150 × 109/L), albumin < 3.5 g/dL (SI unit < 35 g/L), international normalized ratio (INR) > 1.5, total bilirubin > 1.2 mg/dL (SI unit > 20.52 μmol/L), or alpha-fetoprotein (AFP) > 50 ng/mL (SI unit > 180.25 nmol/L). Patients with an elevated indirect bilirubin and known Gilbert's disease can be included if direct bilirubin is within normal limits. Patients with an AFP > 50 ng/mL but ˂ 500 ng/mL can be included if computed tomography (CT) scan or magnetic resonance imaging (MRI) performed within 3 months shows no evidence of hepatocellular carcinoma.
5. Creatinine > 1.2 mg/dL (SI unit > 106.08 μmol/L), creatinine clearance < 50 mL/min (SI unit < 0.83 L/s/m2)
6. Co-infection with hepatitis C virus, human immunodeficiency virus, or hepatitis D virus
7. Evidence or history of hepatocellular carcinoma
8. Malignancy within 5 years prior to Screening, with the exception of specific cancers that are cured by surgical resection (basal cell skin cancer, etc.). Patients under evaluation for possible malignancy are not eligible.
9. Significant cardiovascular, pulmonary, or neurological disease
10. Received solid organ or bone marrow transplant
11. Received within 3 months of Screening or expected to receive prolonged therapy with immunomodulators (e.g., corticosteroids) or biologics (e.g., monoclonal antibody, Interferon)
12. Patients currently taking medication(s) that are transported through organic anion transporting polypeptide 1 including, but not limited to, atazanavir, rifampin, cyclosporine, eltrombopag, gemfibrozil, lopinavir/ritonavir, and saquinavir
13. Use of any herbal medications or supplements during the study period
14. Use of another investigational agent within 3 months of Screening
15. Current alcohol or substance abuse judged by the Investigator to potentially interfere with compliance
16. Females who are pregnant or may wish to become pregnant during the study
17. If the Investigator believes the prospective patient will not be able to comply with the requirements of the protocol and complete the study
18. Any medical condition, in the opinion of the Investigator, that could interfere with evaluation of the study objectives or safety of the patients

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2019-12-21 (Actual); Study Completion 2019-12-21 (Actual)

PRIMARY OUTCOMES:
Change in intra-hepatic immune response | 6 Weeks
  Relative change from Baseline to Week 6 of intra-hepatic immune response (quantitative measurement of 500-600 genes using Nanostring technology) in hepatocytes and liver immune cells derived from the central immunology core biopsy
Change in intra-hepatic anti-viral response | 6 Weeks
  Relative change from Baseline to Week 6 of intra-hepatic anti-viral response (HBV DNA, HBV RNA, HBV core levels, cccDNA and HBsAg levels) using PCR assays in hepatocytes and liver immune cells derived from the intra-hepatic virology biopsy.

SECONDARY OUTCOMES:
Proportion of patients with an adverse event (AE), or a clinically significant clinical laboratory abnormality | 6 weeks
  Proportion of patients during the Baseline to Week 6 inarigivir treatment period with an adverse event (AE), or a clinically significant clinical laboratory abnormality
Correlation of change of intra-hepatic immune markers, serum cytokines and PBMC activation | 6 weeks
  Correlation of change from Baseline to Week 6 of intra-hepatic immune markers, serum cytokines and PBMC activation measured by interferon-stimulated gene (ISG) production
Correlation of change of intra-hepatic antiviral response and serum anti-viral response | 6 weeks
  Correlation of change from Baseline to Week 6 of intra-hepatic antiviral response and serum anti-viral response
Comparison of change of intra-hepatic biomarkers of immune activation | 6 weeks
  Comparison of change in mRNA expression using Nanostring Technology, from Baseline to Week 6 of intra-hepatic biomarkers of immune activation between inarigivir 400 mg per day and 400 mg three times per week
Comparison of change of peripheral biomarkers of immune activation | 6 weeks
  Comparison of change in mRNA expression using Nanostring Technology, from Baseline to Week 6 of intra-hepatic and peripheral biomarkers of immune activation and anti-viral response between inarigivir 400 mg per day and 400 mg three times per week
Comparison of change of anti-viral response | 6 weeks
  Comparison of change in mRNA expression using Nanostring Technology, from Baseline to Week 6 of anti-viral response between inarigivir 400 mg per day and 400 mg three times per week
Characterization of hepatic immune cells | 6 weeks
  Characterization by immuno-phenotyping of hepatic immune cells at Baseline and Week 6. Hepatic immune cells are analyzed and sorted by phenotype using markers of cell activation status through flow cytometry.
Characterization of exhaustion markers | 6 weeks
  Characterization by immuno-phenotyping of exhaustion markers at Baseline and Week 6. Hepatic immune cells are analyzed and sorted by phenotype using markers T cell exhaustion through flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Lim Seng Gee, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore